CLINICAL TRIAL: NCT06751641
Title: A Longitudinal, Multicenter Survey of Adult Participants Enrolled in Decentralized Clinical Trials
Brief Title: Survey of Adult Participants Enrolled in Decentralized Clinical Trials
Acronym: DeCTris
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_LF_DeCTris_01
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Clinical Trial Incorporating Decentralized Elements

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient participating in a clinical trial incorporating decentralized elements. — participating in a clinical trial incorporating decentralized elements.

SUMMARY:
Clinical trials (CTs) have become increasingly complex, requiring significant commitment from participants. Decentralized clinical trials (DCTs) offer an alternative by shifting some activities away from traditional sites to locations like the patient's home. This reduces the burden on participants, improves accessibility, and enhances recruitment and retention rates.

DCTs leverage digital tools such as telemedicine, electronic consent, and wearable devices for data collection. These methods enable fewer site visits, lowering costs and integrating trials more seamlessly into participants' daily routines.

This survey aims to assess the willingness of participants already enrolled in traditional CTs to engage in DCTs. Their prior experience with trial procedures allows them to provide valuable insights into the perceived benefits and feasibility of decentralized elements.

DETAILED DESCRIPTION:
The purpose of this survey is to assess the interest of adults enrolled in a traditional interventional clinical trial involving a drug in participating in a clinical trial incorporating decentralized elements.

ELIGIBILITY:
Inclusion Criteria:

Adults. Patients or healthy volunteers, ambulatory, enrolled in an interventional clinical trial evaluating a drug and receiving the trial treatment(s) either at the investigative site and/or at their place of residence.

Exclusion Criteria:

Individuals who have not expressed their non-opposition to participating in the survey.

Individuals participating in a clinical trial with procedures that are not deemed translatable to decentralized procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population includes adults participating in traditional clinical trials for drugs that could adopt decentralized elements in the future. Eligible participants are patients or healthy volunteers enrolled in interventional trials evaluating one or more drugs, regardless of pathology, receiving treatments at the investigative site and/or their residence.
  Examples include participants in trials for injectable drugs administered in hospitals, such as anticancer agents. However, trials with non-translatable procedures, like those involving critically ill patients in intensive care, are excluded. Anyone meeting these criteria is eligible for the DeCTris survey
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
To assess the willingness of adults already enrolled in an interventional clinical trial involving a drug to participate in a similar trial that incorporates one or more decentralized elements. | 1 day
  "DCT Disposition," is an ordinal variable derived from the DeCTRis self-questionnaire. This scale has five levels, with higher scores indicating a greater willingness to participate in a Decentralized Clinical Trial (DCT). The minimum score is 1, representing the lowest willingness, while the maximum score is 5, indicating the highest willingness to participate in a DCT.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Flet, PharmD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France